CLINICAL TRIAL: NCT05375565
Title: Comparative Effects of Weight Bearing and Non-weight Bearing Exercises on Pain, Range of Motion and Disability in Patients With Total Hip Replacement
Brief Title: Comparative Effects of Weight Bearing and Non-weight Bearing Exercises in Patients With Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0140 Habiba
Record Dates: First submitted 2022-04-26; First posted 2022-05-16 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Total Hip Replacement
Keywords: weight bearing; exercise; hip; pain; replacement; arthroplasty; range of motion
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight bearing exercises (Experimental): weight bearing exercises
  Interventions: Other: weight bearing exercises
- non weight bearing exercises (Experimental): non weight bearing exercises
  Interventions: Other: non weight bearing exercises

INTERVENTIONS:
Other: weight bearing exercises — * Standing knee raise 10 rep x 2sets
  * Standing knee bend 10 rep x 2sets
  * Standing hip extension 10 rep x 2sets
  * Shallow squats 5 rep x 2 sets After 4 week gradually restricting the use of assistive device when patient become able to walk and stand for 10 mins then add stair climbing and descending with a step height not higher than 7 inch.
  The session will be around 45 to 60 minutes on each patient with 2 sessions per week on alternate days to observe the long term effects.
  Arms: weight bearing exercises
Other: non weight bearing exercises — * Seated knee flexion 10 rep x 2sets
  * Seated knee extension 10 rep x2sets
  * Use of stationary bicycle 10 mins
  * Side lying leg lift 10 rep x2sets
  * Straight leg raise 10 rep x 2sets The session will be around 45 to 60 minutes on each patient with 2 sessions per week on alternate days to observe the long term effects.
  Arms: non weight bearing exercises

SUMMARY:
to compare the effects of weight bearing and non-weight bearing exercises on pain, range of motion and disability in patients with total hip replacement

ELIGIBILITY:
Inclusion Criteria:

* unilateral total hip arthroplasty
* posterolateral approach of hip replacement
* patients that were willing to participate
* patients with 2 weeks post-operative history of total hip replacement

Exclusion Criteria:

* History of any systemic pathology
* Individual suffering from congenital hip disease.
* Bilateral total hip arthroplasty
* Evidence of CNS involvement and any other neurological involvement
* Any red flag (malignancies or any kind of tumor
* History of lower extremity fracture.
* Patient having any local or systemic infection of hip joint

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 6 weeks
  NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"
Goniometry | 6 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position
Hip disability and Osteoarthritis Outcome Score (HOOS) | 6 weeks
  A 40 item questionnaire (hip disability and osteoarthritis outcome score, HOOS) was constructed to assess patient-relevant outcomes in five separate subscales (pain, symptoms, activity of daily living, sport and recreation function and hip related quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Lahore General hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wijnen A, Bouma SE, Seeber GH, van der Woude LHV, Bulstra SK, Lazovic D, Stevens M, van den Akker-Scheek I. The therapeutic validity and effectiveness of physiotherapeutic exercise following total hip arthroplasty for osteoarthritis: A systematic review. PLoS One. 2018 Mar 16;13(3):e0194517. doi: 10.1371/journal.pone.0194517. eCollection 2018. PMID 29547670
- [Background] Pozzi F, Madara K, Zeni JA Jr. A SIX-WEEK SUPERVISED EXERCISE AND EDUCATIONAL INTERVENTION AFTER TOTAL HIP ARTHROPLASTY: A CASE SERIES. Int J Sports Phys Ther. 2017 Apr;12(2):259-272. PMID 28515981
- [Background] Mikkelsen LR, Madsen MN, Rathleff MS, Thorborg K, Rossen CB, Kallemose T, Bandholm T. Pragmatic Home-Based Exercise after Total Hip Arthroplasty - Silkeborg: Protocol for a prospective cohort study (PHETHAS-1). F1000Res. 2019 Jun 25;8:965. doi: 10.12688/f1000research.19570.2. eCollection 2019. PMID 31448107
- [Background] Wu JQ, Mao LB, Wu J. Efficacy of exercise for improving functional outcomes for patients undergoing total hip arthroplasty: A meta-analysis. Medicine (Baltimore). 2019 Mar;98(10):e14591. doi: 10.1097/MD.0000000000014591. PMID 30855443
- [Background] Monaghan B, Cunningham P, Harrington P, Hing W, Blake C, O' Dohertya D, Cusack T. Randomised controlled trial to evaluate a physiotherapy-led functional exercise programme after total hip replacement. Physiotherapy. 2017 Sep;103(3):283-288. doi: 10.1016/j.physio.2016.01.003. Epub 2016 Feb 15. PMID 27126617
- [Background] Goh SL, Persson MSM, Stocks J, Hou Y, Welton NJ, Lin J, Hall MC, Doherty M, Zhang W. Relative Efficacy of Different Exercises for Pain, Function, Performance and Quality of Life in Knee and Hip Osteoarthritis: Systematic Review and Network Meta-Analysis. Sports Med. 2019 May;49(5):743-761. doi: 10.1007/s40279-019-01082-0. PMID 30830561
- [Background] Bandholm T, Wainwright TW, Kehlet H. Rehabilitation strategies for optimisation of functional recovery after major joint replacement. J Exp Orthop. 2018 Oct 11;5(1):44. doi: 10.1186/s40634-018-0156-2. PMID 30306337
- [Background] Ackerman IN, Bohensky MA, Zomer E, Tacey M, Gorelik A, Brand CA, de Steiger R. The projected burden of primary total knee and hip replacement for osteoarthritis in Australia to the year 2030. BMC Musculoskelet Disord. 2019 Feb 23;20(1):90. doi: 10.1186/s12891-019-2411-9. PMID 30797228
- [Background] Patel S, Bhanushali Y, Gadhavi B. Effect of Following Physiotherapy on Strength and Range of Motion in Patients with Total Hip Arthroplasty: A Case Series. International Journal of Health Sciences and Research. 2021;11(4):122-32.